CLINICAL TRIAL: NCT02733601
Title: BreCaReAl: Breast Cancers Registry in Algeria
Brief Title: Epidemiology of Breast Cancer in Women Based on Diagnosis Data From Oncologists and Breast Surgeons in Algeria
Acronym: BreCaReAl
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00109
Record Dates: First submitted 2016-03-11; First posted 2016-04-11 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Oncology; Epidemiology; Breast Cancer
Keywords: breast cancer epidemiology algeria registry
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — sodium-iodide symporter; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer Patients: Newly diagnosed with breast cancer all stages confirmed during the study period by an anatomopathologist, defined as a first diagnosis of breast cancer based on anatomopathological results from at least a microbiopsy
  Interventions: Other: NIS (Non Interventional Study) observational study

INTERVENTIONS:
Other: NIS (Non Interventional Study) observational study — NIS observational study : Epidemiologic registry

SUMMARY:
National, prospective, multicentre, non-interventional epidemiological study, conducted among oncologists and breast surgeons in community and university hospitals, from the public sector in Algeria.

The study will collect information on the characteristics, and breast carcinomas patterns of patients whose breast cancer diagnosis was confirmed by an anatomopathologist. The study will be conducted over a representative, but not exhaustive sample of Algerian female patients.

DETAILED DESCRIPTION:
The study consists of:

* Four in-hospital visits (inclusion visit, visit at 3 months, visit at 6 months, visit at 12 months). All patients presenting to their oncologists/breast surgeons during a routine visit and meeting eligibility criteria will be sequentially asked to participate to the study
* In addition to the 4 visits, a phone contact with the patients will be done by the investigator or the CRO (Clinical Research Organization, independent person) or during a routine visit to the investigator, to check the patients' survival every 6 months during 5 years (8 contacts).

Duration of patient recruitment: 6 months from the date of first patient's inclusion.

Duration of patient follow-up: 60 months 3.2 Data Source A comprehensive list of all Algeria hospitals will be used as a data source in the site selection process. The list will be obtained either from the health authority, local scientific societies or professional associations, depending on the local availability of this type of information. All efforts will be made to approach and select sites/physicians.

The oncologist/breast surgeons (investigator) or one of his/her authorised representative in each participating site will complete a CRF (Case Report Form). All data to be collected will be based on the patient's medical file.

The patient will also complete an auto-questionnaire about quality of life at inclusion, 6 and 12 months follow-up.

The CRF will collect all data required for the study and will be transmitted to the project team for analysis following each eligible patient's visit to the investigator.

Data collection should be precise and reliable. The study monitor will verify the authenticity of the data, by matching the CRF with the source documents at the site, and in compliance with the guidelines for good pharmacoepidemiology practices and the recommendations of the Association of French-speaking Epidemiologists (ADELF).

In total, 10 to 15% of the eCRFs (electronic Case Report Form) by site will be verified.

Following the data verification, lists of non-conformity will be generated and transmitted to the study investigators.

The investigator should provide the Sponsor, when requested, all necessary and important data for control. The access to the complete patient's medical file, should be authorised by the investigator, providing that the patient's confidentiality is preserved.

Patients who do not give their written informed consent will only be listed, their data will not be collected on the patient form by the Sponsor.

In case of any particular problem, an audit request can be made.

This study will include representative centres of breast cancer managing departments in each sanitary region defined by the Ministry of health, the investigational centres will propose to all patients whom met eligibility criteria to participate to the study. 1500 patients are expected to be enrolled in the study (incidence study).

Study duration: 66 months

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to participate to the study if they fulfil all of the following criteria:

* Female patients
* Aged 18 years and over
* Newly diagnosed with breast cancer all stages confirmed during the study period by an anatomopathologist, defined as a first diagnosis of breast cancer based on anatomopathological results from at least a microbiopsy
* Provision of subject informed consent.

Exclusion Criteria:

Patients will not be eligible to participate if any of the following criteria are present:

* Informed consent not obtained.
* Patients with a mental or psychological disorder according to their treating clinicians
* Patients participating in an interventional study or already included in the study. A patient could be consulted and treated in two different centres, thus a codification system will be generated to avoid duplicate participation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include representative centres of breast cancer managing departments in each sanitary region defined by the Ministry of health, the investigational centres will propose to all patients whom met eligibility criteria to participate to the study. 1500 patients are expected to be enrolled in the study (incidence study).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-05-29 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Survival status at 05 years (percentage of patients still alive at 05 years) | 60 months
  Survival status at 60 months based on the percentage of patients still alive at 05 years

SECONDARY OUTCOMES:
incidence all cases | 06 months
  Number of new diagnosed cases of breast cancer, all stages combined, by oncologists and breast surgeons, in pre- and post-menopausal women, related to the general female population in Algeria over 06 months of recruitment period.
Incidence by age | 60 months
  Number of new cases diagnosed with breast cancer by age (18 - 20, 20-30, 30 - 40, 40 - 50, 50-60, 60 - 70 and > 70 years old).
Incidence by stage | 60 months
  Number of new diagnosed patients by stage (TNM classification sub population).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Bendib, Oncologist, Principal Investigator — CPMC
Locations (3):
- Algeria (3):
  - Research Site, East of Algeria, East of Algeria
  - Research Site, Middle of Algeria, Middle of Algeria
  - Research Site, Ouest of Algeria/ Oran Region, Ouest of Algeria/ Oran Region

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00109&attachmentIdentifier=f9563843-f638-48ed-928d-facb8ab83479&fileName=BreCaReAl_CSR_Synopsis_Redacted.pdf&versionIdentifier=